CLINICAL TRIAL: NCT02774122
Title: Cochleural Alternating Acoustic Beam Therapy Versus Masking Intervention for Tinnitus: A Randomised Controlled Trial
Brief Title: Cochleural Alternating Acoustic Beam Therapy (CAABT) Versus Masking Intervention for Tinnitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Shu-sheng Gong, director, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 961619
Record Dates: First submitted 2016-05-08; First posted 2016-05-17 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- masking therapy (Active Comparator): Masking intervention was a standard monophone tinnitus masking therapy.
  Interventions: Device: masking therapy
- CAABT (Experimental): CAABT was an innovative tinnitus intervention which based on neural science and cochlear plastic research and aimed to reprogram the central auditory system to neutralize the discordant responses of the dysfunctioning cochlea via acoustic beaming stimuli.
  Interventions: Device: CAABT

INTERVENTIONS:
Device: CAABT — CAABT was an innovative tinnitus intervention which based on neural science and cochlear plastic research and aimed to reprogram the central auditory system to neutralize the discordant responses of the dysfunctioning cochlea via acoustic beaming stimuli.
  Arms: CAABT
Device: masking therapy — Masking intervention was a standard monophone tinnitus masking therapy.
  Arms: masking therapy

SUMMARY:
This study is to compare the effectiveness of CAABT and masking therapy in the management of subjective tinnitus in adults.Half of participants will receive CAABT, while the other half will receive masking therapy.

DETAILED DESCRIPTION:
Masking intervention was a standard monophone tinnitus masking therapy. It was usually a narrow-band noise matched with tinnitus frequency (Tf).

CAABT was an innovative tinnitus intervention which based on neural science and cochlear plastic research and aimed to reprogram the central auditory system to neutralize the discordant responses of the dysfunctioning cochlea via acoustic beaming stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral tinnitus
* Ages between 18-80 years
* Tinnitus undergone for more than 6 months
* Hearing loss of the tinnitus ear not affect communication
* The main tinnitus frequency is less than 8 KHz
* Primary tinnitus

Exclusion Criteria:

* Secondary tinnitus
* Hyperacusis
* Patients were accepting any therapy about tinnitus
* Those who have serious mental illness
* Patients who can't fit the audiological examination and tinnitus tests
* Most of the hearing loss in the middle and severe hearing loss of the tinnitus ear
* Any MRI contraindications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Tinnitus Subjective Measures at 12 weeks: pure tone audiometry | baseline and 12 weeks
Change from Baseline in Tinnitus Subjective Measures at 12 weeks: tinnitus loudness | baseline and 12 weeks
Change from Baseline in Tinnitus Subjective Measures at 12 weeks: minimize masking level | baseline and 12 weeks
Change from Baseline in Tinnitus Subjective Measures at 12 weeks: the Chinese version of Tinnitus Handicap Inventory scale | baseline and 12 weeks
Change from Baseline in Tinnitus Subjective Measures at 12 weeks: the Visual Analog Scale | baseline and 12 weeks

SECONDARY OUTCOMES:
Change from Baseline in Tinnitus Objective Measure at 12 weeks: functional magnetic resonance imaging (fMRI) | baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gong shu-sheng, MD, Study Director — Beijing Friendship Hospital
Locations (1):
- Otorhinolaryngology Head and Neck Surgery department, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
individual participant data(IPD) for all subjective and objective outcome measures will be made available within 6 months of study completion
Supporting Information: Study Protocol
Time Frame: Data will be made available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external Independent Review Panel.

REFERENCES:
- [Result] Cima RF, Maes IH, Joore MA, Scheyen DJ, El Refaie A, Baguley DM, Anteunis LJ, van Breukelen GJ, Vlaeyen JW. Specialised treatment based on cognitive behaviour therapy versus usual care for tinnitus: a randomised controlled trial. Lancet. 2012 May 26;379(9830):1951-9. doi: 10.1016/S0140-6736(12)60469-3. PMID 22633033
- [Derived] Liu C, Zhang J, Qi Z, Yue W, Yuan Y, Jiang T, Zhang S, Zhang S. Therapy effect of cochleural alternating acoustic beam therapy versus traditional sound therapy for managing chronic idiopathic tinnitus patients. Sci Rep. 2024 Mar 11;14(1):5900. doi: 10.1038/s41598-024-55866-0. PMID 38467716
- [Derived] Wei X, Lv H, Wang Z, Liu C, Ren P, Zhang P, Chen Q, Liu Y, Zhao P, Gong S, Yang Z, Wang Z. Neuroanatomical Alterations in Patients With Tinnitus Before and After Sound Therapy: A Voxel-Based Morphometry Study. Front Neurosci. 2020 Sep 8;14:911. doi: 10.3389/fnins.2020.00911. eCollection 2020. PMID 33013302
- [Derived] Liu C, Lv H, Jiang T, Xie J, He L, Wang G, Liu J, Wang Z, Gong S. The Cochleural Alternating Acoustic Beam Therapy (CAABT): A pre-clinical trial. Am J Otolaryngol. 2018 Jul-Aug;39(4):401-409. doi: 10.1016/j.amjoto.2018.04.002. Epub 2018 Apr 3. PMID 29655489